CLINICAL TRIAL: NCT05387902
Title: Short-term Outcomes of Elective High-risk PCI With Extracorporeal Membrane Oxygenation Support: a Single-centre Registry
Status: Completed | Type: Observational
Sponsor: Robert Jan van Geuns (Other)
Responsible Party: Sponsor-Investigator, Robert Jan van Geuns, Prof. dr., Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Other Study IDs: 113382
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO: Patients receiving hemodynamic support with ECMO during high-risk PCI
  Interventions: Device: Extracorporeal Membrane Oxygenation
- ECMO Standby: Patients with ECMO standby during high-risk PCI

INTERVENTIONS:
Device: Extracorporeal Membrane Oxygenation — Patients with high-risk PCI receive mechanical circulatory support with ECMO.
  Groups: ECMO

SUMMARY:
Background Revascularization of complex coronary artery disease, including multivessel coronary artery disease, left main stenosis, bifurcation stenosis and chronic total occlusions (CTO) can be performed by Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Graft (CABG), according to current guidelines.[1] In order to decide whether to revascularize by either CABG or PCI, patient characteristics, the presence of comorbidities, including diabetes, and coronary lesion complexity (e.g. SYNTAX) should be taken into consideration. Because of the ageing population with a higher incidence of comorbidities and higher surgical risk scores, high-risk PCI in complex coronary disease with high risk for periprocedural cardiogenic shock is increasingly performed.[2, 3] Mechanical Circulatory Support (MCS) devices for elective high-risk PCI can provide hemodynamic support, preventing hemodynamic failure during PCI. Several studies are performed using Intra-Aortic Balloon Pump (IABP) and co-axial left cardiac support device (Impella device (Abiomed, Danvers, USA)), showing no clear benefits in patients with high-risk PCI.[4-6] Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO) is a recent addition to mechanical support options, providing more extensive hemodynamic support in patients with potential or ongoing failure of circulation. This concept is already demonstrated in the setting of Extracorporeal Cardiopulmonary Resuscitation (ECPR).[7, 8] ECMO has the additional benefits of right ventricular unloading and blood oxygenation as opposed to IABP and Impella.[9] Our experience with fully percutaneous VA-ECMO in cardiogenic shock and for ECPR combined with the experience for Transcatheter Aortic Valve Replacement (TAVR) with local anaesthesia and mild sedation resulted in the selection of VA-ECMO as our preferred method in high risk PCI. Studies investigating the use of VA-ECMO support during high-risk PCI are however limited.[10-13]

Objective The aim of this study is to provide additional data concerning the short-term outcomes of elective high-risk PCI with VA-ECMO in a single PCI centre.

Methods Design We will perform a single-centre, retrospective registry, using data collected from medical records of included patients.

Inclusion criteria

* Patients older than 18 years, who underwent high-risk PCI with VA-ECMO support.
* The use of mechanical circulatory support (MCS) is indicated by HeartTeam based on patient and lesion characteristics described in the expert consensus on the use of MCS Devices for high-risk PCI. [14]

Exclusion criteria

• Non-elective PCI with VA-ECMO support, primarily applied for cardiogenic shock or ECPR.

Study Procedures All patients older than 18 years who underwent high-risk PCI with VA-ECMO support will be included in the registry. Baseline patient and angiographic characteristics, ECMO characteristics and short-term outcomes, described in the paragraph 'Study Endpoints and Definitions' will be collected from medical records.

The Dutch Act on Medical Research involving Human Subjects (WMO) does not apply to this study, because of the retrospective design of the study using only medical records and consequently patients are not subjected to additional procedures. Therefore, no written informed consent will be obtained from patients or legal representatives as well.

Data Collection All data will be collected in a cloud-based electronic case report form (eCRF, Castor Electronic Data Capture), which will be developed and managed by investigators in the Radboudumc. Only members of the study team will have access to the patient eCRFs and will be allowed to enter data in the system. The study team exists of the investigators mentioned earlier. The study team will collect the data from medical records and enter the data in Castor. All patient data will be encoded. Only the investigators involved will have access to the patient identification key.

Study Endpoints and Definitions Successful revascularization is defined as final residual stenosis <50% with a TIMI flow grade 3, achieved in at least one of the target vessels. Procedural success is defined as angiographic success without the occurrence of peri-procedural MACE, including death and myocardial infarction (MI). Additionally, MACE will be assessed during hospital stay and within 60-days follow-up after discharge and defined as a composite of death, MI, Target Vessel Revascularization (TVR) by PCI or CABG and clinical bleeding, assessed by the Bleeding Academic Research Consortium (BARC) scale. Bleeding complications of type 2 and higher are included.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, who underwent high-risk PCI with VA-ECMO support.
* The use of mechanical circulatory support (MCS) is indicated by HeartTeam based on patient and lesion characteristics described in the expert consensus on the use of MCS Devices for high-risk PCI.

Exclusion Criteria:

- Non-elective PCI with VA-ECMO support, primarily applied for cardiogenic shock or ECPR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients older than 18 years who are undergoing a high-risk PCI with VA-ECMO support, indicated by HeartTeam consensus based on patient and lesion characteristics, as described by the expert consensus. If a non-elective PCI with VA-ECMO support, primarily applied for cardiogenic shock or ECPR, is performed, patients are not eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | from PCI procedure up to hospital discharge, an average of 7 days
  Composite of death, MI, Target Vessel Revascularization (TVR) by PCI or CABG and clinical bleeding, assessed by the Bleeding Academic Research Consortium (BARC) scale
Major Adverse Cardiac Events | within 60 days after discharge
  Composite of death, MI, Target Vessel Revascularization (TVR) by PCI or CABG

SECONDARY OUTCOMES:
Succesful Revascularization | During PCI Procedure
  Final residual stenosis <50% with a TIMI flow grade 3, achieved in at least one of the target vessels
Procedural Success | During PCI Procedure
  Angiographic success without the occurrence of peri-procedural MACE, including death and myocardial infarction (MI)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan M van Geuns, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon request, data supporting the findings and conclusion of this study will be made available by the PI.

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Valgimigli M, Tebaldi M, Borghesi M, Vranckx P, Campo G, Tumscitz C, Cangiano E, Minarelli M, Scalone A, Cavazza C, Marchesini J, Parrinello G; PRODIGY Investigators. Two-year outcomes after first- or second-generation drug-eluting or bare-metal stent implantation in all-comer patients undergoing percutaneous coronary intervention: a pre-specified analysis from the PRODIGY study (PROlonging Dual Antiplatelet Treatment After Grading stent-induced Intimal hyperplasia studY). JACC Cardiovasc Interv. 2014 Jan;7(1):20-8. doi: 10.1016/j.jcin.2013.09.008. Epub 2013 Dec 11. PMID 24332420
- [Background] Waldo SW, Secemsky EA, O'Brien C, Kennedy KF, Pomerantsev E, Sundt TM 3rd, McNulty EJ, Scirica BM, Yeh RW. Surgical ineligibility and mortality among patients with unprotected left main or multivessel coronary artery disease undergoing percutaneous coronary intervention. Circulation. 2014 Dec 23;130(25):2295-301. doi: 10.1161/CIRCULATIONAHA.114.011541. Epub 2014 Nov 12. PMID 25391519
- [Background] Perera D, Stables R, Thomas M, Booth J, Pitt M, Blackman D, de Belder A, Redwood S; BCIS-1 Investigators. Elective intra-aortic balloon counterpulsation during high-risk percutaneous coronary intervention: a randomized controlled trial. JAMA. 2010 Aug 25;304(8):867-74. doi: 10.1001/jama.2010.1190. PMID 20736470
- [Background] Perera D, Stables R, Clayton T, De Silva K, Lumley M, Clack L, Thomas M, Redwood S; BCIS-1 Investigators. Long-term mortality data from the balloon pump-assisted coronary intervention study (BCIS-1): a randomized, controlled trial of elective balloon counterpulsation during high-risk percutaneous coronary intervention. Circulation. 2013 Jan 15;127(2):207-12. doi: 10.1161/CIRCULATIONAHA.112.132209. Epub 2012 Dec 6. PMID 23224207
- [Background] Henriques JP, Remmelink M, Baan J Jr, van der Schaaf RJ, Vis MM, Koch KT, Scholten EW, de Mol BA, Tijssen JG, Piek JJ, de Winter RJ. Safety and feasibility of elective high-risk percutaneous coronary intervention procedures with left ventricular support of the Impella Recover LP 2.5. Am J Cardiol. 2006 Apr 1;97(7):990-2. doi: 10.1016/j.amjcard.2005.10.037. Epub 2006 Feb 13. PMID 16563902
- [Background] Bougouin W, Dumas F, Lamhaut L, Marijon E, Carli P, Combes A, Pirracchio R, Aissaoui N, Karam N, Deye N, Sideris G, Beganton F, Jost D, Cariou A, Jouven X; Sudden Death Expertise Center investigators. Extracorporeal cardiopulmonary resuscitation in out-of-hospital cardiac arrest: a registry study. Eur Heart J. 2020 Jun 1;41(21):1961-1971. doi: 10.1093/eurheartj/ehz753. PMID 31670793
- [Background] Yannopoulos D, Bartos J, Raveendran G, Walser E, Connett J, Murray TA, Collins G, Zhang L, Kalra R, Kosmopoulos M, John R, Shaffer A, Frascone RJ, Wesley K, Conterato M, Biros M, Tolar J, Aufderheide TP. Advanced reperfusion strategies for patients with out-of-hospital cardiac arrest and refractory ventricular fibrillation (ARREST): a phase 2, single centre, open-label, randomised controlled trial. Lancet. 2020 Dec 5;396(10265):1807-1816. doi: 10.1016/S0140-6736(20)32338-2. Epub 2020 Nov 13. PMID 33197396
- [Background] Spiro J, Doshi SN. Use of left ventricular support devices during acute coronary syndrome and percutaneous coronary intervention. Curr Cardiol Rep. 2014 Dec;16(12):544. doi: 10.1007/s11886-014-0544-x. PMID 25326728
- [Background] Vainer J, van Ommen V, Maessen J, Geskes G, Lamerichs L, Waltenberger J. Elective high-risk percutaneous coronary interventions supported by extracorporeal life support. Am J Cardiol. 2007 Mar 15;99(6):771-3. doi: 10.1016/j.amjcard.2006.10.034. Epub 2007 Jan 22. PMID 17350362
- [Background] Shaukat A, Hryniewicz-Czeneszew K, Sun B, Mudy K, Wilson K, Tajti P, Stanberry L, Garberich R, Sandoval Y, Burke MN, Chavez I, Gossl M, Henry T, Lips D, Mooney M, Poulose A, Sorajja P, Traverse J, Wang Y, Bradley S, Brilakis ES. Outcomes of Extracorporeal Membrane Oxygenation Support for Complex High-Risk Elective Percutaneous Coronary Interventions: A Single-Center Experience and Review of the Literature. J Invasive Cardiol. 2018 Dec;30(12):456-460. PMID 30504514
- [Background] van den Brink FS, Meijers TA, Hofma SH, van Boven AJ, Nap A, Vonk A, Symersky P, Sjauw KD, Knaapen P. Prophylactic veno-arterial extracorporeal membrane oxygenation in patients undergoing high-risk percutaneous coronary intervention. Neth Heart J. 2020 Mar;28(3):139-144. doi: 10.1007/s12471-019-01350-8. PMID 31782108
- [Background] Tomasello SD, Boukhris M, Ganyukov V, Galassi AR, Shukevich D, Haes B, Kochergin N, Tarasov R, Popov V, Barbarash L. Outcome of extracorporeal membrane oxygenation support for complex high-risk elective percutaneous coronary interventions: A single-center experience. Heart Lung. 2015 Jul-Aug;44(4):309-13. doi: 10.1016/j.hrtlng.2015.03.005. Epub 2015 Apr 23. PMID 25913808
- [Background] Rihal CS, Naidu SS, Givertz MM, Szeto WY, Burke JA, Kapur NK, Kern M, Garratt KN, Goldstein JA, Dimas V, Tu T; Society for Cardiovascular Angiography and Interventions (SCAI), Heart Failure Society of America (HFSA), Society of Thoracic Surgeons (STS), American Heart Association (AHA), and American College of Cardiology (ACC). 2015 SCAI/ACC/HFSA/STS Clinical Expert Consensus Statement on the Use of Percutaneous Mechanical Circulatory Support Devices in Cardiovascular Care: Endorsed by the American Heart Association, the Cardiological Society of India, and Sociedad Latino Americana de Cardiologia Intervencionista; Affirmation of Value by the Canadian Association of Interventional Cardiology-Association Canadienne de Cardiologie d'intervention. J Am Coll Cardiol. 2015 May 19;65(19):2140-1. doi: 10.1016/j.jacc.2015.02.043. Epub 2015 Apr 7. No abstract available. PMID 25861962
- [Derived] Griffioen AM, Van Den Oord SCH, Van Wely MH, Swart GC, Van Wetten HB, Danse PW, Damman P, Van Royen N, Van Geuns RJM. Short-Term Outcomes of Elective High-Risk PCI with Extracorporeal Membrane Oxygenation Support: A Single-Centre Registry. J Interv Cardiol. 2022 Sep 16;2022:7245384. doi: 10.1155/2022/7245384. eCollection 2022. PMID 36189196